CLINICAL TRIAL: NCT04363476
Title: Preventing Post-traumatic Osteoarthritis and Other Health Consequences Following Knee Joint Injury: A Pilot Randomized Controlled Trial
Brief Title: Preventing Knee Osteoarthritis Through Exercise and Education Following Knee Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sport Injury Prevention Research Centre (Other)
Responsible Party: Principal Investigator, Carolyn Emery, Professor, Sport Injury Prevention Research Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REB19-0276
Record Dates: First submitted 2020-04-01; First posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Osteoarthritis Knees Both Post-Traumatic
Keywords: osteoarthritis; prevention; exercise
MeSH Terms: conditions — Osteoarthritis; Motor Activity

STUDY DESIGN:
Intervention Model Description: Step-wedge design with two parallel arms
Who Masked: Investigator, Outcomes Assessor
Masking Description: Research assistants performing testing and data entry and the investigators performing analysis will be blinded throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 8-week exercise and education intervention. Two 60-minute physiotherapist-lead group exercise classes with education incorporated will be delivered weekly for 8 weeks (16 classes). In addition, participants will complete a 30-minute home exercise session once a week for 8-weeks (8 sessions). After the intervention, the group will enter a 16-week maintenance stage. During maintenance, a 30-minute home exercise program is completed twice a week.
  Interventions: Other: SHRED Osteoarthritis program
- Control (Other): The control group will not receive an intervention during the first 8-weeks of the study. Being a step-wedge design, this group will receive the same 8-week exercise and education intervention later, after the intervention group has completed the intervention and the post-intervention testing. After the control group has completed the 8-week intervention, they will enter an 8-week maintenance stage. During maintenance, a 30-minute home exercise program is completed twice a week.
  Interventions: Other: SHRED Osteoarthritis program

INTERVENTIONS:
Other: SHRED Osteoarthritis program — Combined exercise and education intervention

SUMMARY:
This study evaluates the preliminary efficacy of an 8-week exercise and education intervention on musculoskeletal health of young adults with a previous sport-related knee injury that are at high risk of post-traumatic osteoarthritis. In addition, the purpose of this pilot randomized controlled trial is to determine the feasibility of the study methods and procedures to inform the design of a future randomized controlled trial.

DETAILED DESCRIPTION:
PURPOSE

The purpose of this study is to determine the preliminary efficacy of an 8-week exercise and education intervention on musculoskeletal health of young adults with a previous sport-related knee injury that are at high risk of post-traumatic osteoarthritis. In addition, the purpose is to determine the feasibility of the study methods and procedures. In addition, the longitudinal changes in health-related factors in participants who are recruited from a previous cohort study will be described, as well as the estimated cost of healthcare utilization during one year in a population of young adults with history of sport-related knee injury.

METHODS

Study design and participants

This is a pilot randomized controlled trial stepped-wedge design. Participants will include 40 men and women, age 21 to 33 years, who sustained a physician-confirmed youth (≤ 18 years of age) sport-related intra-articular knee injury 5 to 16 years ago.

Participants will be randomly assigned to the intervention group (n=20) or the control group (n=20) in permuted blocks of varying size and stratified during randomization by sex. To ensure allocation concealment, the trial biostatistician, who is not involved in participant recruitment or baseline testing, will generate the randomization sequence. After the participant has been tested at baseline, the study physiotherapist will open the envelope and informed the participant about allocation to intervention or control group. If a participant expresses that they are unable to participate in the group they were allocated to, they will not be excluded from this pilot study. Instead, they are permitted to participate in the group that is suitable to them. The number of these cases will be recorded and reported.

All participants will undergo baseline testing at the same time. Intervention group will then complete the 8-week intervention, while the control group will not begin the intervention until 8 weeks after their baseline measurements. Intervention group will complete a 16-week maintenance period while control group will complete eight weeks of maintenance. All participants will undergo functional (i.e. balance and strength) tests, body composition measurements, 7-day physical activity monitoring and fill self-report tools (i.e. Knee Injury and Osteoarthritis Outcome Score, knee self-efficacy) at four time points: baseline, 8-weeks, 16-weeks and 24-weeks.

Experimental Intervention: the SHRED Osteoarthritis program

Exercise Component:

Previous research on the effects of neuromuscular training after knee injuries and on patients with knee OA, research on neuromuscular control, exercise training principles and the research group's clinical experience were considered when designing the exercise component of the SHRED Osteoarthritis program. The SHRED Osteoarthritis program consists of an an 8-minute warm-up, 42-minute circuit training through seven exercise stations, 5 minutes of specialized skill and control exercises and 5-minute cool down inclusive of flexibility exercises.

The SHRED Osteoarthritis program will be delivered through two 60-minute group exercise classes per week for 8 weeks (16 classes). In addition, participants will complete a 30-minute home exercise session once a week (8 sessions). The SHRED Osteoarthritis exercise classes will be lead by a study physiotherapist assisted by kinesiologists, kinesiology students or physiotherapy students with a supervision rate of one instructor for every four participants.

The 30-minute home exercise sessions will consist of a warm-up (8 min) and four exercises from the SHRED Osteoarthritis program. The physiotherapist leading the SHRED Osteoarthritis classes will assign specific exercises to each participant, based on individual needs and the program will be revised weekly.

Education Component:

Patient education is embedded into the 16, one-hour supervised group exercise classes. Education components will include the causes and course of knee pain, identification of a flare-up, management and first aid for self-management of knee pain or flare-ups, appropriate imaging, exercise progression and treatment options (conservative vs. surgical). This content was built from clinical practice guidelines, expert recommendations, patient interviews and theoretical frameworks that outline patient needs, modifiable risk factors, proposed change objects and performance objectives.

Maintenance Component:

After the 8-week intervention has been completed, participants will enter a maintenance stage. During this time (16 weeks for intervention group, 8 weeks for control group), the participants will be asked to complete an individualized home exercise program twice a week. During the maintenance period, participants have the opportunity to contact the study physiotherapist via phone or email to discuss their progression and possible changes to their program. In addition, drop-in times will be available twice a week. During these times, participants can come to discuss their program with the study physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Sustained a physician-confirmed intra-articular sport-related knee injury in age 18 years or younger

Exclusion Criteria:

* Injury or a flare-up at the time of recruitment, which makes the individual unable to participate in more than two exercises in the exercise program
* Pregnancy
* Any contraindication to exercise
* Lower extremity surgery within the last 6 months
* Already attending structured supervised exercise or other treatment to improve knee function
* Not available to participate in the weekly exercise classes

Ages: 21 Years to 33 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-04 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Knee Extension Strength | Baseline, 8-weeks, 16-weeks and 24-weeks
  Normalized knee extension strength will be assessed using hand-held isometric dynamometry. The peak isometric strength (N) from the three trials will be recorded for both legs. The peak isometric strength scores are converted to torque values (Nm; force x distance between joint line and dynamometer position) and normalized to body weight (Nm/kg). The mean value of the three trials will be calculated.
Participation Rate | Duration of the 8-week intervention for both study groups (week 1 to 8 for intervention group, week 9 to 16 for control group.
  Attendance in the group exercise classes and completion of the home exercise sessions will be recorded. Participation rate for the two study groups (intervention/control) will be calculated as the proportion of completed group exercise classes and home exercise sessions out of the total possible group exercise classes and home exercise sessions over the 8-week intervention.

SECONDARY OUTCOMES:
Retention Rate | The duration of the study (weeks 1-24), will be calculated in the end.
  Retention rate will be described as the proportion of randomized participants retained the end of the study out of the total number of randomized participants.
Joint-Specific Adverse Events | The duration of the study (weeks 1-24)
  The number of joint-specific adverse events will be recorded. Joint-specific adverse events are determined as participant not attending an exercise session and/or ceasing participation due to increased pain or problems in the index knee and self-reported pain greater than 5 on a scale of 0 to 10 scale after an exercise session.
Self-reported Pain Before and After Exercise | Duration of the 8-week intervention for both study groups (week 1 to 8 for intervention group, week 9 to 16 for control group.
  Self-reported pain will be measured on a scale of 0 to 10. Pain will be monitored before class, in the end of the class, and 24 hours after class. Participants will record the pain score in their individual training diary before and after class. To record pain score 24 hours after class, a text message or an email (depending on participant's preference) containing a link to record the pain score will be sent using research electronic data capture (REDCap) software.
Major and Minor Adverse Events | The duration of the study (weeks 1-24)
  Major and minor adverse events will be reported following the CONSORT extension statement for harms-reporting in randomized clinical trials. Major events are defined as death or hospitalization within trial care or 3 hours after. Minor events are defined as other unwanted outcomes that requires clinician attention.
Program Progression Achieved | Duration of the 8-week intervention for both study groups (week 1 to 8 for intervention group, week 9 to 16 for control group.
  Participants' progression during the 8-week exercise intervention will be recorded for each exercise station as the level of progression achieved in the end of the intervention. Four levels of progression are used (1-4).
Observed Exercise Fidelity | Duration of the 8-week intervention for both study groups (week 1 to 8 for intervention group, week 9 to 16 for control group.
  Observed exercise fidelity will be assessed using a checklist consisting of essential criteria for each exercise variation. Exercise fidelity will be expressed as percentage of exercise criteria achieved and will be recorded for each exercise as well as the complete program.
Measured Exercise Fidelity | Duration of the 8-week intervention for both study groups (week 1 to 8 for intervention group, week 9 to 16 for control group.
  Exercise fidelity during the group exercise sessions will be measured for all participants using inertial measurement units (IMUs). Measured exercise fidelity will be determined using a binary support vector machine classification model built to determine exercise fidelity for each exercise. Measured exercise fidelity will be expressed as percentage of exercise criteria achieved.
Average Heart Rate | Each supervised group exercise class (twice a week for 8 weeks)
  Average heart rate (pbm) during the group exercise class measured using a heart rate monitor with a chest strap during the group exercise classes.
Maximum Heart Rate | Each supervised group exercise class (twice a week for 8 weeks)
  Maximum heart rate (pbm) during the group exercise class measured using a heart rate monitor with a chest strap during the group exercise classes.
Time at Heart Rate Zone of 50 to 60 percent of HRmax | Each supervised group exercise class (twice a week for 8 weeks)
  Time spent (as minutes) on heart rate zone of 50 to 60 percent of age-predicted maximum heart rate during the group exercise classes.
Time at Heart Rate Zone of 61 to 70 percent of HRmax | Each supervised group exercise class (twice a week for 8 weeks)
  Time spent (as minutes) on heart rate zone of 61 to 70 percent of age-predicted maximum heart rate during the group exercise classes.
Time at Heart Rate Zone of 71 to 80 percent of HRmax | Each supervised group exercise class (twice a week for 8 weeks)
  Time spent (as minutes) on heart rate zone of 71 to 80 percent of age-predicted maximum heart rate during the group exercise classes.
Time at Heart Rate Zone of 81 to 90 percent of HRmax | Each supervised group exercise class (twice a week for 8 weeks)
  Time spent (as minutes) on heart rate zone of 81 to 90 percent of age-predicted maximum heart rate during the group exercise classes.
Time at Heart Rate Zone of >90 percent of HRmax | Each supervised group exercise class (twice a week for 8 weeks)
  Time spent (as minutes) on heart rate zone of >90 percent of age-predicted maximum heart rate during the group exercise classes.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Baseline, 8-weeks, 16-weeks and 24-weeks
  The KOOS consists of 42 items in five subscales: pain, other symptoms, function in daily living, function in sport and recreation, and knee related quality of life. Each item is scored on a 5-point Likert scale ranging from no problems to extreme problems. The subscale scores are summed, and the total score is transformed to a 0-100 scale with higher scores indicating better function.
Health-related Quality of Life (EQ-5D-5L) | Baseline, 8-weeks, 16-weeks and 24-weeks
  The Canadian algorithm will be used to calculate the EuroQol 5 Dimension Questionnaire (EQ-5D-5L) score. The value set range for Canadians -0.148 (worst health status, worse than dead) to 0.949 (best health status).
Knee Self-efficacy (K-SES) | Baseline, 8-weeks, 16-weeks and 24-weeks
  The K-SES covers four domains of self-efficacy: 1) daily activities (seven items), 2) sport and leisure activities (five items), 3) physical activities (six items), and 4) knee function in the future (four items). The response to the 22 items is given using an 11-grade Likert scale, ranging from 0 (not at all certain about the task) to 10 (very certain about the task). The sum of item scores is calculated and divided by the number of items. The total score is transformed to a 0-100 scale with higher score indicating better self-efficacy.
Intermittent and Constant Osteoarthritis Pain (ICOAP) | Baseline, 8-weeks, 16-weeks and 24-weeks
  The ICOAP consists of 11 items forming two subscales. Each item was scored on a 5-point Likert scale ranging from no pain to high (disability-severely limiting) pain. Sub-scale scores will be summed and the total score transformed to a 1-100 scale (higher scores indicating poorer outcome).
Tampa Scale for Kinesiophobia (TSK) | Baseline, 8-weeks, 16-weeks and 24-weeks
  The TSK consists of 17 items. Each item is scored on a 4-point Likert scale, ranging from 1 'strongly disagree' to 4 'strongly agree'. The range of total score is from 17 to 68. Higher scores indicate higher levels of kinesiophobia.
Healthcare Utilization | Baseline
  Healthcare utilization (i.e., visits to healthcare professionals, treatments, tests and services) will be based on participant self-report, on an item-by-item basis, for the 1-year period preceding testing. Current (2018) unit costs and rules from the Alberta Health Services Calgary Zone will be applied to value the health care system resources used by participants.
Knee Flexion Strength | Baseline, 8-weeks, 16-weeks and 24-weeks
  Normalized knee flexion strength will be assessed at using hand-held isometric dynamometry. The peak isometric strength (N) scores are converted to torque values (Nm; force x distance between joint line and dynamometer position) and normalized to body weight (Nm/kg).
Hip Abduction Strength | Baseline, 8-weeks, 16-weeks and 24-weeks
  Normalized hip abduction strength will be assessed at using hand-held isometric dynamometry. The peak isometric strength (N) scores are converted to torque values (Nm; force x distance between joint line and dynamometer position) and normalized to body weight (Nm/kg).
Hip Adduction Strength | Baseline, 8-weeks, 16-weeks and 24-weeks
  Normalized hip adduction strength will be assessed at using hand-held isometric dynamometry. The peak isometric strength (N) scores are converted to torque values (Nm; force x distance between joint line and dynamometer position) and normalized to body weight (Nm/kg).
Triple Single-Leg Hop | Baseline, 8-weeks, 16-weeks and 24-weeks
  Each participant will perform two trials of three consecutive single-leg hops with the goal of jumping as far as possible. Both legs will be tested (starting with the non-injured leg), and the maximum distance (cm) from the two trials normalized for leg length will be recorded for each leg.
Single-Leg Hop for Distance | Baseline, 8-weeks, 16-weeks and 24-weeks
  The test will be performed until three successful trials have been recorded for both legs. Hop distance is measured in centimeters (cm) from the toe at the push-off to the heel where the subject landed. The maximum distance (cm) from the three trials normalized for leg length will be recorded for each leg.
Y-Balance Test | Baseline, 8-weeks, 16-weeks and 24-weeks
  Three complete rounds on each leg will be completed with three reaching distances. The maximal reach distance (cm) at the point where the most distal part of the foot reaches is measured and normalized for lower extremity length. The normalised composite score will be calculated.
Moderate-to-vigorous Physical Activity | Baseline, 8-weeks, 16-weeks and 24-weeks
  To determine the average daily minutes of moderate-to-vigorous PA (MVPA), all participants will wear a waist-mounted accelerometer device for seven days. Minutes of MVPA will be calculated based on activity corresponding to moderate activity 3-6 metabolic equivalents of task (MET) and vigorous activity >6 MET. A log will be used to record non-wear time (i.e. water-based activities) and activities with very limited vertical movement (i.e. spin class and cycling).
Asymmetries in Jumping Performance | Baseline, 8-weeks, 16-weeks and 24-weeks
  Five inertial measurement units (Blue Trident IMU, Vicon Motion Systems Inc) will be attached to the body at the lower back, near the centre of mass and on the distal anteromedial aspect of each tibia. During the data collection participants will perform ten maximal countermovement jumps and ten maximal squat jumps with 30 second rest between jumps. Asymmetry in each phase will be reported as the difference between the left and right limb impulses divided by the maximum limb impulse and expressed as a percentage.
Fat mass index | Baseline, 8-weeks, 16-weeks and 24-weeks
  Dual-energy x-ray absorptiometry (DXA) scanner will be used to capture whole body composition scans. Fat mass index will be calculated as fat mass relative to stature squared (kg/m^2).
Body mass index | Baseline, 8-weeks, 16-weeks and 24-weeks
  Body mass index (BMI; kg/m^2) will be calculated from height (to the nearest 0.1 cm; shoes removed) and weight (to the nearest 0.1 kg) assessed using a medical scale and stadiometer.
Lean mass index | Baseline, 8-weeks, 16-weeks and 24-weeks
  Dual-energy x-ray absorptiometry (DXA) scanner will be used to capture whole body composition scans. Lean mass index will be calculated as lean mass relative to stature squared (kg/m2).
Number of Exercise Sessions Completed during the Maintenance Stage | Maintenance stage (weeks 9 to 24 for intervention group, weeks 17 to 24 for control group)
  The total number of times the home exercise session was completed during the maintenance stage will be recorded.
Weekly Time Spent Completing the Program during the Maintenance Stage | Maintenance stage (weeks 9 to 24 for intervention group, weeks 17 to 24 for control group)
  The weekly minutes spent completing the home exercise sessions during the maintenance stage will be recorded.
Joint-specific Adverse Events during the Maintenance Stage | Maintenance stage (weeks 9 to 24 for intervention group, weeks 17 to 24 for control group)
  The number of joint-specific adverse events will be recorded during the maintenance stage. Joint-specific adverse events are determined as participant not attending an exercise session and/or ceasing participation due to increased pain or problems in the index knee and self-reported pain greater than 5 on a scale of 0 to 10 scale after an exercise session.
Consultations with the Study Physiotherapist during the Maintenance Stage | Maintenance stage (weeks 9 to 24 for intervention group, weeks 17 to 24 for control group)
  Total number of times the participants consulted the study physiotherapist during the maintenance stage to discuss their home exercise program.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn A Emery, PT, PhD, Principal Investigator — Sport Injury Prevention Research Centre, University of Calgary
Locations (1):
- University of Calgary Sport Injury Prevention Research Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Relph N, Greaves H, Armstrong R, Prior TD, Spencer S, Griffiths IB, Dey P, Langley B. Running shoes for preventing lower limb running injuries in adults. Cochrane Database Syst Rev. 2022 Aug 22;8(8):CD013368. doi: 10.1002/14651858.CD013368.pub2. PMID 35993829